CLINICAL TRIAL: NCT02497157
Title: Phase II Trial of FOLFOXIRI + Bevacizumab in Patients With Untreated Metastatic Colorectal Cancer
Brief Title: Bevacizumab + Triplet Treatment for Untreated With Chemotherapy Metastatic Colorectal Cancer
Acronym: BeTRI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Hiroshima Prefectural Hospital (Unknown); National Hospital Organization Shikoku Cancer Center (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRICC1414; UMIN000017102 (Other: UMIN-CTR)
Record Dates: First submitted 2015-06-25; First posted 2015-07-14 (Estimated); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Metastatic Colorectal Cancer
Keywords: bevacizumab; oxaliplatin; irinotecan; hydrochloride hydrate; fluorouracil; levofolinate calcium
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; Irinotecan; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): Patients receive FOLFOXIRI plus bevacizumab [oxaliplatin (L-OHP): 85 mg/sq.m., irinotecan hydrochloride hydrate (CPT-11): 165 mg/sq.m., continuous intravenous infusion of fluorouracil (CIV 5-FU): 3,200 mg/sq.m., Levofolinate calcium (l-LV): 200 mg/sq.m., bevacizumab: 5 mg/kg]. The treatment will be repeated every 2 weeks, for up to 12 cycles, unless the disease progression, unacceptable toxicity, tumor resection or consent withdrawal.
  Interventions: Drug: Oxaliplatin (L-OHP); Drug: Irinotecan hydrochloride hydrate (CPT-11); Drug: Continuous intravenous infusion of fluorouracil (CIV 5-FU); Drug: Levofolinate calcium (l-LV); Drug: Bevacizumab (Bmab)

INTERVENTIONS:
Drug: Oxaliplatin (L-OHP)
Drug: Irinotecan hydrochloride hydrate (CPT-11)
Drug: Continuous intravenous infusion of fluorouracil (CIV 5-FU)
Drug: Levofolinate calcium (l-LV)
Drug: Bevacizumab (Bmab)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of fluorouracil (5-FU), levofolinate calcium (l-LV), oxaliplatin (L-OHP) and irinotecan hydrochloride hydrate (CPT-11) (FOLFOXIRI) plus bevacizumab in untreated metastatic colorectal cancer patients who harbor Uridine diphosphate (UDP)-glucuronosyl transferase 1A1 (UGT1A1) *1/*1, *1/*6 or *1/*28.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the colon or rectum.
2. Unresectable or recurrent colorectal cancer patient.
3. One or more measurable lesion in RECIST ver.1.1 criteria.
4. No prior chemotherapy, immunotherapy, and radiotherapy.
5. Life expectancy at least 3 months.
6. Patients who harbor UGT1A1*1/*1, *1/*6 or *1/*28.
7. The Eastern Cooperative Oncology Group (ECOG) performance status of =<1.
8. Vital organ functions (listed below) are preserved within 14 days prior to entry.

   White blood cell count (WBC): >= 3,000 per cubic millimeter Neu: >= 1,500 per cubic millimeter Platelet count (PLT): >= 100,000 per cubic millimeter Aspartate aminotransferase (AST/GOT) and alanine aminotransferase (ALT/GPT): <= 100 IU/L, <= 150 IU/L in cases with liver metastasis T-bil: <= 1.5 mg/dL Serum creatinine: <= 1.50 mg/dL Proteinuria: <= 1+ Prothrombin time-international normalized ratio (PT-INR): < 1.5
9. Written informed consent.

Exclusion Criteria:

1. Vermiform appendix cancer and anal canal cancer.
2. Administration of blood products/ granulocyte-colony stimulating factor (G-CSF), and blood transfusion within 14 days prior to enrollment.
3. Synchronous multiple malignancy or metachronous multiple malignancy less than 5 years disease free interval.
4. Hepatitis B virus antigen (HBs-Ag)(+), or hepatitis C virus antibody (HCV-Ab)(+).
5. History of severe allergy.
6. Sensory alteration or paresthesia interfering with function.
7. Prior radiotherapy for ilium and abdomen.
8. Infectious disease.
9. Uncontrolled diarrhea.
10. Ileus or bowel obstruction.
11. Interstitial lung disease or pulmonary fibrosis.
12. Malignant coelomic fluid required drainage.
13. Administration of atazanavir sulfate.
14. Heart disease to be clinically problem.
15. Major surgical procedure or intestinal resection within 28 days prior to enrollment or colostomy within 14 days prior to enrollment.
16. Known brain metastasis or strongly suspected of brain metastasis.
17. History of a thromboembolic disease.
18. Receiving anti-platelet drugs.
19. Poorly controlled gastrointestinal ulcer.
20. History of intestinal perforation within the past 12 months.
21. Poorly controlled hypertension.
22. Poorly controlled diabetes mellitus.
23. Severe mental disorders.
24. Women who are pregnant or nursing, men and women who wish to conceive a child or with no intention to contraception.
25. Any other cases who are regarded as inadequate for study enrollment by investigators.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2015-05-21 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Response rate (RR) by response evaluation criteria in solid tumors (RECIST v1.1) | Up to 18 months
  RR will be calculated as the ratio of the number of eligible patients who experienced a confirmed Complete response(CR) or Partial response(PR) by RECIST v1.1.

SECONDARY OUTCOMES:
Time to treatment failure (TTF) | Up to 18 months
  TTF is defined as the time from date of starting treatment until date of treatment discontinuation, the first documented progression or death from any cause, whichever comes first.
Progression-free survival (PFS) | Up to 3 years
  PFS is defined as the time from date of starting treatment until date of the first documented progression or death from any cause, whichever comes first.
Overall survival (OS) | Up to 3 years
  OS is defined as the time from date of starting treatment until date of death from any cause.
R0 resection rate | Up to 18 months
  R0 resection rate will be calculated as the ratio of the number of eligible patients who experienced a complete (R0) resection.
Relative dose intensity (RDI) | Up to 18 months
  RDI will be calculated as the ratio of actual delivered dose intensity in comparison with planned dose intensity. Dose intensity (DI) is defined as the amount of drug delivered per unit time, expressed in mg/m2/week.
Incidence of adverse events | Up to 3 years

OTHER OUTCOMES:
Early tumor shrinkage (ETS) rates in 8 weeks after starting the treatment, evaluated by RECIST v1.1 | Baseline (week 0), week 8
  ETS will be calculated as the ratio of the number of eligible patients who experienced a 20% or more tumor shrinkage at week 8 compared with baseline.
Deepness of response (DoR) | Up to 3 years
  DoR will be calculated as the median of the maximum tumor shrinkage rates.

CONTACTS AND LOCATIONS:
Overall Officials: Katsunori Shinozaki, MD, Ph.D., Principal Investigator — Hiroshima Prefectural Hospital; Tomohiro Nishina, MD, Ph.D., Principal Investigator — National Hospital Organization Shikoku Cancer Center
Locations (7):
- Japan (7):
  - Matsuyama Red Cross Hospital, Matsuyama, Ehime
  - Kagawa University Hospital, Kita-gun, Miki-cho, Kagawa-ken
  - Kawasaki Medical School Hospital, Kurashiki, Okayama-ken
  - Okayama Saiseikai General Hospital, Okayama, Okayama-ken
  - Okayama University Hospital, Okayama, Okayama-ken
  - Okayama Rosai Hospital, Okayama, Okayama-ken
  - Tokushima Red Cross Hospital, Komatsushimachō, Tokushima